CLINICAL TRIAL: NCT06270628
Title: Demonstrating the (Cost-)Effectiveness of a Personalized Live-remote Exercise Intervention for Cancer Survivors Using a Super Umbrella Randomized Controlled Trial: the LION RCT
Brief Title: Personalized Live-remote Exercise Training for Cancer Survivors
Acronym: LION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: German Cancer Research Center (Other); German Sport University Cologne (DSHS), Cologne, Germany (Unknown); Cabrini Health (CAB), Malvern, Australia (Unknown); Karolinska Institute (KI), Stockholm, Sweden (Unknown); Netherlands Cancer Institute (NKI), Amsterdam, The Netherlands (Unknown); Heidelberg University Clinic and National Center for Tumor Diseases, Heidelberg, Germany (Unknown); Fundacion Onkologikao (ONK), San Sebastian, Spain (Unknown); Associação de Investigação e Cuidados de Suporte em Oncologia (AISCO), Nova de Gaia, Portugal (Unknown)
Responsible Party: Principal Investigator, Dr. Anne May, Prof. Dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL85029.018.23
Record Dates: First submitted 2024-01-15; First posted 2024-02-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Neoplasms
Keywords: cancer survivors; exercise; live remote; personalized exercise training
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: RCT with two study arms: exercise group and wait list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Participants will be offered three live-remote exercise training sessions per week. Each participant in the trial will be provided with the base module twice a week, which will involve a personalized training intensity. This module aims at targeting the participants' HRQOL, which is the first primary endpoint of the trial. Additionally, each participant will receive one out of four specific modules once a week to address their individual main side-effect (based on shared decision-making (SDM)) (second primary outcome). The intervention also includes an educational component about exercise and cancer.
  Interventions: Behavioral: Exercise group
- Wait list control group (No Intervention): Regular care The control group will receive the same exercise program after the 12 weeks intervention period

INTERVENTIONS:
Behavioral: Exercise group — Live-remote exercise sessions, personalized to the patients main side-effect
  Arms: Exercise group

SUMMARY:
Background

Many people with cancer face ongoing problems from their disease and treatments, like fatigue, reduced physical fitness, feeling anxious or down, and neuropathy. While exercise might help with these problems, most studies did not focus on tailoring exercise to address these specific complaints. Exercise programs under supervision (like with a trainer) seem to work better, but barriers for following such sessions are travel distance and time. Therefore, following an exercise program at home with a trainer guiding via video (live-remote) might be a good solution. But, it is unclear how effective this remote exercise program is for cancer patients.

Goal of the study:

The main goal of this study is to assess the effectiveness of a personalized, live-remote exercise intervention for cancer survivors on quality of life and the patients' main complaint. The four complaints tackled in this study are: 1) fatigue, 2) reduced physical functioning, 3) anxiety and/or depressive symptoms, and 4) neuropathy.

Design of the study

In the LION study, 350 cancer patients will be randomly divided into the exercise group or control group. These patients all have at least one of these complaints: 1) fatigue, 2) reduced physical functioning, 3) anxiety and/or depressive symptoms, and/or 4) neuropathy. Patients cannot participate in the study if they are already very active.

The exercise group will start a 12-week exercise program right away, and the other group will wait for 12 weeks before starting. The exercise program consists of three sessions per week. Two sessions per week include aerobic training and strength training. These sessions will be followed by all patients; and aim to improve fitness and strength. The third session specifically aims at improvement of the main complaint, for example fatigue.

Participants will get an app and a fitness tracker to help them stay on track with their exercises. Furthermore, patients get information on the effects of exercise for cancer patients and why exercise is important for specific complaints.

Measurements

The main outcomes of this study are quality of life and the main side-effect of the patient. Other measurements include all kind of patient reported outcomes (like sleep problems and pain), physical fitness, muscle strength, balance, anthropometrics, and (inflammatory) markers in blood.

Conclusion:

This study investigates if personalized exercises done at home, with video guidance, can make cancer survivors feel better and manage their side effects more effectively.

DETAILED DESCRIPTION:
SUMMARY

Rationale:

Many cancer patients suffer from long-term treatment-related side-effects like fatigue, low physical functioning, anxiety and/or depressive symptoms, and chemotherapy-induced peripheral neuropathy (CIPN). There is convincing evidence on the beneficial effects of general exercise interventions on these side-effects. However, studies to date generally fail to specifically screen for (long-term) side-effects at baseline and tailor the intervention to these specific side-effects, although larger exercise effects are observed in patients with a high symptom burden at baseline (e.g., with higher levels of fatigue). Larger effects of exercise are also observed for supervised exercise compared to unsupervised exercise. However, two of the most common barriers for attending and complying with supervised exercise are travel distance and time. An effective approach might be to provide live-remote supervision for exercise interventions. In this scenario, patients can receive guidance from a certified exercise specialist through a video-conferencing platform such as Zoom, while performing exercises within the comfort of their own homes. Currently, the effectiveness of live-remote exercise in cancer patients has not been established.

Objective:

The primary objective of the LION RCT is to assess the (cost-)effectiveness of a personalized, live-remote exercise intervention for cancer survivors on Health-Related Quality of Life (HRQOL) and the participants' main, self-reported side-effect. The four side-effects targeted in this study are: 1) fatigue, 2) perceived low physical functioning in daily life, 3) anxiety and/or depressive symptoms, and 4) CIPN.

Study design:

The LION RCT is a randomized controlled trial with two study arms: an exercise group (12 weeks) and a wait list control group. A super umbrella design will be used, allowing us to evaluate four exercise modalities (i.e., exercise modules based on participants' main side-effect) in a wide variety of cancer survivors.

Study population:

For this study, 350 adult cancer survivors treated with systemic chemotherapy (≥ 12 weeks to 1 year after completion of primary treatment of invasive cancer with curative intent) will be recruited independent of their primary cancer diagnosis. Participants will have reported at least one of the following side-effects: fatigue, low physical functioning in daily life, anxiety and/or depressive symptoms, CIPN. Additionally, participants need to be relatively physically inactive, i.e., perform ≤210 minutes/week of moderate-to-vigorous leisure and sports activities.

Intervention:

The intervention consists of three live-remote exercise sessions per week. Participants randomized to the exercise group receive the intervention after the baseline visit and the wait list control participants after the 12-week follow-up visit. A modular approach will be used to tailor the intervention to each participant's specific main side-effect. Each participant will receive the same base module (twice a week) to address HRQOL and in addition one out of four specific modules (once a week) addressing their individual main side-effect. In addition to the live-remote training, participants will be provided with the LION app and an activity tracker (Fitbit) at the start of the intervention to support exercise beyond the supervised program, during holidays and after the end of the intervention. In addition to exercise, the intervention also has an educational component including information about general effects of exercise for cancer patients and why exercise is important for specific side-effects. We consider the provision of such education as an integral part of adequate exercise programming.

After the intervention period of 12 weeks, we follow the patients until 36 weeks. In this follow-up period, also two sub studies take place:

1. Sensor-based guidance sub study (only control patients from Cologne)
2. Live-remote physical fitness and function testing (in all control patients; all sites)

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, a subject must be:

* 18 years of age or older
* Diagnosed with any type of invasive cancer and have received systemic chemotherapy as part of their primary cancer treatment
* Within the timeframe of 12 weeks to 1 year after the completion of their primary cancer treatment with curative intent. Primary treatment, in this context, includes surgery, radiotherapy, and/or chemotherapy. For patients undergoing endocrine, targeted, or immunotherapy, their treatment must not be scheduled to be discontinued within the next 6 months.
* No evidence of distant metastatic disease (i.e., no diagnosis of metastatic disease in the regular clinical trajectory)
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2
* Presence of at least one of the following side-effects: fatigue (measured using EORTC QLQ-C30 fatigue symptom scale, score >39), perceived low physical functioning in daily life (measured using EORTC QLQ-C30 physical functioning scale, score <83), anxiety or depressive symptoms (measured using PHQ-ADS > 20), and/or CIPN (measured using 2 PRO-CTCAE items, score >0) for patients who received neurotoxic chemotherapy. Cut-off values are based on established thresholds.19-21
* Access to good quality and stable internet connection to access the live-remote training sessions.
* Able and willing to perform the exercise program and wear the activity tracker at least one week after T0 and before T2, T4, and T5 measurements and during training and online assessment sessions.
* Able to read, speak and understand the main country language.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Too physically active (i.e., >210 minutes/week of self-reported moderate-to-vigorous or leisure and sports activities; this threshold has also been used in other exercise RCTs, such as PREFERABLE-EFFECT22, and fits activity levels of all participating countries) or participation in an exercise program comparable to the LION exercise program.
* Following, or planned to follow, a structured psychological intervention during the intervention period, i.e., cognitive behavioral therapy, or unstable on psychotropic medication
* Participated in the intervention group of an exercise study during cancer treatment
* Inability to complete the testing or training sessions or any other contraindications for exercise as determined by the treating physician, including:
* Severe neurologic or cardiac impairment according to ACSM criteria
* Uncontrolled severe respiratory insufficiency or dependence on oxygen suppletion in rest or during exercise
* Uncontrolled pain All these exclusion criteria are formulated to ensure safe participation in the LION exercise program
* Any circumstances that would impede ability to give informed consent or adherence to study requirements as determined by the treating physician
* More than 1 week not able to attend training sessions during the LION intervention period

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | Week 0 - Week 12
  Measured with the summary scale of the EORTC QLQ-C30; min 0- max 100 points; higher scores mean better quality of life
A standardized symptom score, per patient, based on the individual patient's main side-effect defined at baseline | Week 0 - Week 12
  Side-effect 1: Fatigue measured with EORTC QLQ-FA12. According to a standardization procedure the symptom score of all patients will be combined into one symptom score..
A standardized symptom score, per patient, based on the individual patient's main side-effect defined at baseline | Week 0 - Week 12
  Side-effect 2: Anxiety and depressive symptoms measured with Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). According to a standardization procedure the symptom score of all patients will be combined into one symptom score.
A standardized symptom score, per patient, based on the individual patient's main side-effect defined at baseline | Week 0 - Week 12
  Side-effect 3: Physical functioning measured with EORTC QLQ-C30 physical function scale According to a standardization procedure the symptom score of all patients will be combined into one symptom score.
A standardized symptom score, per patient, based on the individual patient's main side-effect defined at baseline | Week 0 - Week 12
  Side-effect 4: CPIN measured with EORTC QLQ-CPIN20. According to a standardization procedure the symptom score of all patients will be combined into one symptom score.

SECONDARY OUTCOMES:
Health-related quality of life | Week 0 - Week 36
  Domains of the EORTC QLQ-C30 (except summary score)
Fatigue | Week 0 - Week 36
  Cancer-Related fatigue measured with the EORTC-FA12
Anxiety and Depression | Week 0 - Week 36
  Anxiety and depressive symptoms measured with the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS)
CIPN_1 | Week 0 - Week 36
  Chemotherapy-induced peripheral neuropathy measured with EORTC QLQ-CIPN-20
CIPN_2 | Week 0 - Week 36
  2 items of the Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Sleep | 0-36 weeks
  Pittsburgh Sleep Quality Index (PSQI)
Pain prevalence and type | Week 0 - Week 36
  EORTC QLQ-SURV100
Cognitive problems | Week 0 - Week 36
  Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog)
Work limitations | Week 0 - Week 36
  Work Limitations Questionnaire (WLQ)
Body image | Week 0 - Week 36
  Body Image Scale (BIS)
Fear of cancer recurrence | 0-36 weeks
  EORTC QLQ-surv100
Habitual physical activity | Week 0 - Week 36
  Modified Godin-Shephard Leisure-Time Physical Activity Questionnaire
Aerobic capacity on bike | Week 0 - Week 24
  Steep ramp test
Aerobic capacity on step | Week 0 - Week 24
  Chester step test
Handgrip strength | Week 0 - Week 24
  Handgrip test
Upper body muscle strength | Week 0 - Week 24
  Chest press
Lower body muscle strength | 0-24 weeks
  Leg press
Sit to stand test | Week 0 - Week 24
  30 sec sit to stand test- function test
Physical function | Week 0 - Week 24
  Time Up and Go (TUG) test
Balance | Week 0 - Week 24
  Single leg stance test with open and closed eyes
Physical activity | 0-36 weeks
  Measured with an activity tracker (Fitbit)
Blood pressure | 0-24 weeks
  Measured twice with blood pressure device
Resting heart rate | Week 0 - Week 24
  Measured with blood pressure device
Weight | Week 0 - Week 24
  Weight. in KG
Height | Week 0 - Week 24
  Height in cm
Waist circumference | Week 0 - Week 24
  Waist circumference in cm
Hip circumference | Week 0 - Week 24
  Hip circumference in cm
Body composition | Week 0 - Week 24
  Fat mass and fat free mass with bio-impedance - three centers
Inflammatory state | 0-12 weeks
  The specific inflammatory markers (e.g., cytokines, interleukins) will be decided at the time-point of analyses to be able to include factors according to up-to-date insights and use state-of the art platforms; we will for example use the Olink PEA platform (Oncology and Inflammation Array)
Growth factors | 0-12 weeks
  The specific growth factors will be decided at the time-point of analyses to be able to include factors according to up-to-date insights and use state-of the art platforms ; we will for example use the Olink PEA platform (Oncology and Inflammation Array)
CRP | Week 0 - Week 12
  Blood cell count
Hemoglobin | 0-12 weeks
  Blood cell count
Leucocyte counts | 0-12 weeks
  Blood cell count
Quality-adjusted life years | Week 0 - Week 36
  EuroQol-5D-5L
Health-care, patient and family costs | Week 0 - Week 36
  Modified Medical Consumption Questionnaire (iMCQ)
Productivity losses | Week 0 - Week 36
  Modified Productivity Cost Questionnaire (iPCQ)
Exercise-related (serious) adverse events | Week 0 - Week 36
  Via CASTOR app before and after each session; asked at and at the study visits.

OTHER OUTCOMES:
Participants experience of sensor-based guidance | Week 12- Week 24
  Questionnaires - substudy control patients Cologne
Trainer experience of sensor-based guidance | Week 12- Week 24
  Questionnaires - substudy control patients Cologne
Compliance sensor-based guidance | Week 12- Week 24
  % of sessions that patients wear the sensor - substudy control patients Cologne
Technical feasibility of sensor-based guidance | Week 12- Week 24
  % of successful live transfer of sensor data - substudy control patients Cologne
Aerobic capacity | Week 12- Week 24
  Chester Step test - substudy live-remote testing
Upper body muscle strength | Week 12- Week 24
  Push-up test - substudy live-remote testing
Lower body muscle strength | Week 12- Week 24
  30 sec sit-to stand test - substudy live-remote testing
Core muscle strength | Week 12- Week 24
  Plank position holding time - substudy live-remote testing
Physical functioning | Week 12- Week 24
  Time Up and Go (TUG) test - substudy live-remote testing
Balance | Week 12- Week 24
  Single leg stance test with open and closed eyes - substudy live-remote testing
Socio-demographics | baseline
  Self-designed questionnaire
Self-efficacy | baseline
  General Self-Efficacy Scale
Social Support | baseline
  Index of Sojourner Social Support (ISSS)
Medical history | baseline
  Interview
Concomitant diseases | Week 0- Week 36
  Interview
Cancer + concomitant medication | Week 0- Week 36
  Interview
Cancer characteristics | baseline
  Interview
Cancer treatment history | baseline
  Interview

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study analyses by the study team, the data will be anonymized and made available for sharing requests.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the study analyses by the study team (TBD).
Access Criteria: TBD in the DMP.

REFERENCES:
- [Derived] Hiensch AE, Muller J, Zopf EM, Schmidt ME, Monninkhof EM, Trevaskis M, Belloso J, Clauss D, Gunasekara N, Joaquim A, Viamonte S, Schumann M, Heinrich L, Kias A, Binyam D, van de Poll L, Buffart LM, Aaronson NK, van der Wall E, Campbell A, Wiskemann J, Rundqvist H, Alves AJ, Urruticoechea A, Bloch W, Stuiver MM, Wengstrom Y, Steindorf K, May AM. Effects of personalized live-remote exercise for individuals living beyond primary curative cancer treatment: study protocol for a multinational, super umbrella randomized controlled trial (LION-RCT). Trials. 2025 Nov 24;26(1):540. doi: 10.1186/s13063-025-09263-1. PMID 41287048
- See also: study website — https://www.preferable2.eu